CLINICAL TRIAL: NCT05655143
Title: Effects of Balance Training on Corticospinal Excitability in People With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Ryan McCann, Assistant Professor, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1957702-4
Record Dates: First submitted 2022-12-06; First posted 2022-12-19 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Training (Experimental)
  Interventions: Behavioral: Balance training
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Balance training — Participants will undergo a 4-week balance training protocol modified from that described previously.
  Participants will undergo supervised exercise three times per week for approximately 30 minutes per session. The exercise consists of single-leg balance training, hop to stabilization, and hop to stabilization plus reaching activities as presented in Figure 1. Particularly, the levels of difficulty will be progressed with visual conditions (eyes open and eyes closed), time (sec), and base of support (floor and foam pad) while hopping distance (inches) for single-leg and hopping activities, respectively. These activities will be progressed in difficulty as participants become proficient at the task.
  Arms: Balance Training

SUMMARY:
Ankle sprains are prevalent and debilitating injuries in daily living and sports activities. The emergency room annually cares for over 206,000 patients with lateral ankle sprain in the United States, resulting in over $12,000 of health care cost per injury. Although many rehabilitation techniques for ankle sprains have been implemented, up to 40% of individuals with ankle sprains experience residual symptoms including recurrent sprain, episodes of ankle joint "giving way," and feelings of instability, which collectively define chronic ankle instability (CAI). Individuals with CAI commonly exhibit neuromuscular dysfunction with reduced motor control due to decreased sensory input to the central nervous system (CNS) after the initial injury. As a result, the CNS sends altered motor signals to lower extremity muscles. These CNS changes contribute to various neuromuscular impairments in CAI patients, the most common of which is reduced balance performance.

Neural stimulation techniques, such as the Hoffman reflex (H-reflex) and transcranial magnetic stimulation (TMS) have been used to directly assess changes in the CNS. One of the most consistently identified CNS changes in individuals with CAI is reduced ability to modulate spinal reflex excitability and corticospinal excitability of the calf muscle when transitioning from simpler to more complex balance conditions. Neural excitability refers to the ability of the central nervous system to elicit skeletal muscle contractions. That is, the spinal reflex excitability and corticospinal excitability can be described as the ability to contract muscle conducted by the spine and brain, respectively. Typically, healthy individuals modulate or quiet down their spinal reflexes and rely more on the corticospinal excitability during more demanding balance tasks. However, evidence indicates that the individuals with CAI are unable to modulate spinal reflexes and shift control to brain, leading to reduced balance performance. Given that the calf muscle plays a crucial role in balance, improving proper supraspinal and spinal reflexive control of the calf muscle is imperative to balance maintenance of individuals with CAI.

To improve balance function for those with CAI, many balance training programs have been implemented to improve static and dynamic stability and proprioception for those with CAI. The majority of findings indicate that balance training can be effective in preventing initial and recurrent ankle sprains. However, it is unclear if common balance training methods can restore the function of the CNS in those with CAI. Therefore, the purpose of this study is to determine the effects of balance training on the calf muscle spinal-reflexive excitability modulation, corticospinal excitability, and balance performance in individuals with CAI. The rationale for this study is that patients with CAI require effective rehabilitation that can restore their neurosignature and improve balance ability.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 to 40 years old
* A previous history of a significant ankle sprain that caused pain and swelling (initial ankle sprain is required to occur at least 12 months prior to study enrollment; the most recent ankle sprain must occur at least 3 months prior to study enrollment)
* At least two recurrent episodes of "giving way," "feeling of instability," or repeated ankle sprains in the six months before the study enrollment
* Scored ≥5 on the Ankle Instability Instrument (AII), >10 on the Identification of Functional Ankle Instability (IdFAI), and <24 on the Cumberland Ankle Instability Tool (CAIT).

Exclusion Criteria:

* Participants should not have any kind of neurological, vestibular, respiratory, or heart disorders, previous surgery, smoke or history of illicit drug use, or be pregnant.
* history of heart disease
* history of stroke
* cardiac pacemaker or implanted cardiac defibrillator
* history of migraines or severe headaches
* history of cancer in brain or leg muscles
* diagnosed psychiatric disorder
* intracranial metallic clips
* currently pregnant or breastfeeding
* taking pain relieving, neuroinhibitory, or stimulating medication within 7 days prior to testing
* metal implants anywhere in the head, neck, or shoulders (excluding dental work)
* personal or familial history of seizures or epilepsy
* ocular foreign objects or cochlear implants
* implanted brain stimulators
* aneurysm clips
* implanted medication pump
* intra- cardiac lines
* history of or is currently abusing illicit drugs or alcohol or is currently withdrawing from any substance
* history of serious head injury or increased intracranial pressure that would keep participants from participating in this study.
* smokers
* diagnosed with a neurologic disorder (e.g., Parkinson's disease, multiple sclerosis, or stroke)
* cognitive status that does not allow the individual to consistently comprehend and repeat back directions regarding the details of the study
* diabetes
* fibromyalgia
* peripheral neuropathy (i.e., numbness, tingling, or loss of sensation in the hands or feet)
* history of acute head or lower extremity injury within 3 months prior to testing
* any history of lower extremity fracture or surgery
* currently using any of the following types of medications:

  * Pain relief medications: common examples include Aspirin, Acetaminophen (Tylenol), Morphine, Tramadol (Ultram), Oxycodone (Percocet), Hydrocodone (Vicodin)
  * Neuroinhibitory medications: common examples include Alprazolam (Xanax), Diazepam (Valium), Clonazepam (Klonopin), Baclofen (Lioresal),

    o These medications are commonly used to treat anxiety and seizures.
  * Stimulating medications: common examples include Methylphenidate (Ritalin), Amphetamine (Adderall), Caffeine

    o These medications are commonly used to treat ADD and narcolepsy.
  * Tricyclic antidepressants: common examples include Amitriptyline, Amoxapine, Desipramine (Norpramin), Doxepin, Imipramine (Tofranil), Nortriptyline (Pamelor), Protriptyline (Vivactil), Trimipramine (Surmontil)

    o These medications are commonly used to treat depression, agoraphobia with panic attacks, obsessive compulsive disorder, chronic pain, and migraine headaches.
  * Neuroleptic (antipsychotic) medications: common examples include Chlorpromazine (Thorazine), Loxapine (Loxitane), Clozapine (Clozaril) o These medications are commonly used to treat psychoses and schizophrenia.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Active Motor Threshold | 1 year
  Transcranial magnetic stimulation will be delivered to the primary motor cortex of each participant using a Magstim Super RAPID2 PLUS1 System. A Double Cone Coil will be positioned over the primary motor cortex's approximated representation of the soleus to deliver single-pulse stimulations. From the output of the soleus MEP, the spot that generates the highest electromyographic (EMG) amplitudes with consistency will be identified as the "hotspot". To acquire the active motor threshold (AMT), the average peak amplitude of the background EMG signal will be collected while participants conduct the single-leg balance without magnetic stimulus. AMT will be defined as the lowest stimulator intensity needed to generate 4/8 stimulations with soleus EMG activity 2 standard deviations above baseline EMG data.
Motor Evoked Potential | 1 year
  After testing active motor threshold (AMT) 8 stimulations at intensities of 100% and 120% of AMT will be delivered using single-pulse stimulations over the soleus "hot spot." The electromyographic activity of the soleus from each stimulation will be recorded as the motor evoked potential (MEP).
Corticosilent Period | 1 year
  From the same stimulations used to test motor evoked potential (MEP), we measure corticosilent period (CSP) as the time from the end of MEP to a return of baseline electromyographic activity of the soleus.
Spinal Reflexive Excitability Modulation | 1 year
  Spinal reflexive excitability modulation will be measured while the participants are in the prone position and a single-leg stance. As a first step, the spinal reflexive excitability during prone and single-leg balance will be determined using a ratio of the Hoffmann-reflex (H-reflex) to the muscle response (M-wave) (H:M). H-reflex and M-wave will be elicited by BIOPAC stimulator module with a 2mm shield disk stimulating electrode attached to the popliteal fossa to stimulate the tibial nerve. The stimulation will be progressively increased with 0.2V until the maximal H-reflex and M-wave are obtained. Five the maximal H-reflex and M-wave will be recorded to calculate the H:M ratio. The following formula will be employed to calculate the modulation of H-reflex:
  (Prone-Single leg standing H:M Ratio)/(Prone H:M ratio)×100
Balance function | 1 year
  Balance performance will be measured via a force platform (AccuSway Plus, AMTI, Watertown, MA, USA) by doing a single-leg standing. The force platform will be connected to the Balance Clinic software (AMTI, Watertown, MA, USA) to acquire the center of pressure (COP) data. Balance function testing will include two visual conditions (Eyes open vs Eyes closed) while participants maintain single-leg balance on the involved limb. Each condition will be conducted three 20-second trials. Averaged COP path length, area, and maximum velocity in anterior-posterior and medial-lateral directions will be utilized for the final data analysis. Rest intervals of 1 minute will be provided between each condition. Furthermore, subjects will be protected by the primary investigator to prevent falling from the base of supports.
  3)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Brain Research and Rehabilitation, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No